CLINICAL TRIAL: NCT05232669
Title: COcoa Supplement and Multivitamin Outcomes Study (COSMOS): Effects on Falls and Physical Performance
Brief Title: COcoa Supplement and Multivitamin Outcomes Study: Effects on Falls and Physical Performance
Acronym: COSMOS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Meryl LeBoff, Principal Investigator, Brigham and Women's Hospital
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: 2021P003714; 2021A008958 (Other: MGB)
Record Dates: First submitted 2022-01-31; First posted 2022-02-10 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Fall; Physical Performance; Fracture
MeSH Terms: conditions — Fractures, Bone | interventions — Chocolate; Geritol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cocoa extract + multivitamin (Active Comparator)
  Interventions: Dietary Supplement: Cocoa extract; Dietary Supplement: Multivitamin
- Cocoa extract + multivitamin placebo (Active Comparator)
  Interventions: Dietary Supplement: Cocoa extract; Dietary Supplement: Multivitamin placebo
- Cocoa extract placebo + multivitamin (Active Comparator)
  Interventions: Dietary Supplement: Cocoa extract placebo; Dietary Supplement: Multivitamin
- Cocoa extract placebo + multivitamin placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Cocoa extract placebo; Dietary Supplement: Multivitamin placebo

INTERVENTIONS:
Dietary Supplement: Cocoa extract — 2 capsules each day containing a total of 500 mg cocoa flavanols, including 80 mg (-)-epicatechin, and 50 mg theobromine
  Arms: Cocoa extract + multivitamin; Cocoa extract + multivitamin placebo
Dietary Supplement: Cocoa extract placebo — Cocoa extract placebo
  Arms: Cocoa extract placebo + multivitamin; Cocoa extract placebo + multivitamin placebo
Dietary Supplement: Multivitamin — Multivitamin
  Arms: Cocoa extract + multivitamin; Cocoa extract placebo + multivitamin
Dietary Supplement: Multivitamin placebo — Multivitamin placebo
  Arms: Cocoa extract + multivitamin placebo; Cocoa extract placebo + multivitamin placebo

SUMMARY:
The COcoa Supplement and Multivitamin Outcomes Study (COSMOS; NCT02422745) is a randomized clinical trial of cocoa extract supplement (containing a total of 500 mg/d flavanols, including 80 mg. (-)-epicatechins), and a standard multivitamin supplement to reduce the risk of cardiovascular disease and cancer among men aged 60 years and older and women aged 65 years and older. This ancillary study is being conducted among participants in COSMOS and will examine whether the cocoa extract supplement or the multivitamin supplement improve musculoskeletal health and prevent falls and declining physical performance in the increasing number of older adults in the U.S. with potential for clinical and public health benefits.

ELIGIBILITY:
Participants in COSMOS (NCT02422745) who meet the following criteria are eligible to participate in this ancillary study:

1. Participants who reported an injurious fall resulting in healthcare utilization (visit to a healthcare provider or hospital)
2. Participants who reported recurrent falls (2 or more falls per year)

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21442 (Actual)
Dates: Start 2021-05-15 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Injurious falls resulting in healthcare utilization (visit to a healthcare provider or hospital) | 5 years
Recurrent falls (2 or more falls per year) | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Meryl S LeBoff, MD, Principal Investigator — Brigham and Women's Hospital; Carolyn Crandall, MD, MS, Principal Investigator — University of California, Los Angeles
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] LeBoff MS, Chou SH, Ratliff KA, Cook NR, Clar A, Holman B, Copeland T, Smith DC, Rist PM, Manson JE, Sesso HD, Crandall CJ. Rationale and design of an ancillary study evaluating the effects of the cocoa flavanol and/or multivitamin interventions on falls and physical performance outcomes in the COcoa Supplement and Multivitamin Outcomes Study (COSMOS). Contemp Clin Trials. 2023 Feb;125:107078. doi: 10.1016/j.cct.2023.107078. Epub 2023 Jan 6. PMID 36621596
- See also: COSMOS Trial Website — http://www.cosmostrial.org/